CLINICAL TRIAL: NCT02735434
Title: Internet-delivered Acceptance and Commitment Therapy for Patients With Health Anxiety: a Randomized Controlled Trial
Brief Title: Internet-delivered Acceptance and Commitment Therapy for Patients With Health Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09032016
Record Dates: First submitted 2016-04-01; First posted 2016-04-12 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2017-03

CONDITIONS: Hypochondriasis
Keywords: Health anxiety; illness anxiety disorder; ACT; internet
MeSH Terms: conditions — Hypochondriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Internet-based ACT (Experimental): Brief clinical psychiatric assessment to determine eligibility (video-based).
  Interventions: Behavioral: Internet-based ACT
- Internet-based discussion forum (Active Comparator): Brief clinical psychiatric assessment to determine eligibility (video-based).
  Interventions: Other: Internet-based discussion forum

INTERVENTIONS:
Behavioral: Internet-based ACT — The guided internet program consists of 7 modules activated consecutively over a period of 12 weeks. The content is written psycho education, patient videos, audio-exercises and behavioural exposure exercises. The program is therapist-guided; hence all patients will receive support from primarily the same therapist during the 12 weeks.
  Arms: Internet-based ACT
Other: Internet-based discussion forum — The online discussion forum consists of 7 themes touching upon the impact of health anxiety and the patients own coping strategies. The themes are activated consecutively over a period of 12 weeks. The discussion forum is text-based, and only patients will participate in the discussion. The written discussions will be reviewed by a professional for ethical reasons. The discussion forum aims to control for the effect of attention and contacts to the health care system. After 9 months patients in the discussion forum are offered active treatment, but not as part of the research project.
  Arms: Internet-based discussion forum

SUMMARY:
Health anxiety is a prevalent, disabling disorder associated with extensive health care expenditures. The lack of easily accessible, evidence-based psychological treatment combined with delayed diagnostic recognition constitute barriers to receiving treatment.

Aim

1. To develop an internet-delivered treatment program, based on 'Acceptance and Commitment Therapy' (ACT), for patients with health anxiety.
2. To test the feasibility and effectiveness of the treatment programme in a randomized, controlled trial, comparing the treatment with an active control condition.

Methods 150 patients aged 18 years and older can self-refer through a web-page to apply for participation. Before inclusion patients will undergo a video-diagnostic interview. Patients are randomly assigned to 12 weeks of either, 1) active treatment: consisting of internet-based ACT (iACT) with 7 therapist-guided modules of self-help text, exercises, patient videos and audio-files, or 2) active control condition: consisting of an internet-based discussion forum (iFORUM) with 7 topics of discussion.

All patients will complete self-report questionnaires at baseline, before randomization, at 4 and 8 weeks into treatment, after end of treatment, and at 6-month follow-up.

DETAILED DESCRIPTION:
Severe health anxiety (illness anxiety disorder) or hypochondriasis, according to the psychiatric classification system ICD-10, is characterized by preoccupation with fear of having a serious illness, which interferes with daily functions and persists despite medical reassurance. Clinical significant health anxiety is prevalent in primary care with 0.8-9.5%, and has a lifetime prevalence of 5.7% in the general population. It is a disabling disorder, associated with extensive use of health care services and occupational disability.

Earlier, health anxiety has been considered a chronic disease with poor treatment outcomes. A recent review found effect of both medicine and psychotherapy, but patients may prefer psychotherapeutic treatments. Despite the high prevalence, health anxiety is rarely diagnosed within primary care, and there is limited access to evidence-based treatment for health anxiety.

An easily accessible, evidence-based treatment is needed for this debilitating condition.

Internet-based treatment is a new approach where patients receive access to a guided self-help program. A meta-analysis has shown equal treatment effects of internet-based treatment compared to "face-to-face" treatment for depressive- and anxiety disorders. Internet-based cognitive behavioral therapy for health anxiety has shown to be cost-effective. ACT is a new effective generation of cognitive-behavioral therapy, with an emphasis on acceptance and value-based exposure that has shown good results for treating health anxiety in a group setting. Internet-based Cognitive behavioral therapy (CBT) for health anxiety has shown promising results but low treatment completion. This may be due to the comprehensive treatment modules and the text-based format. ACT is an experiential behavioral therapy, and aims to activate patients with exercises, videos, audio-files and less text material.

Most persons with health anxiety have high health care expenditure. However, some patients with health anxiety avoid contact to the health care system, and may not receive proper treatment. Patient self-referral is a new approach that may facilitate access to treatment.

Aim

1. To develop an internet-delivered treatment program for patients suffering from health anxiety based on ACT.
2. To test the feasibility and effectiveness of the treatment programme in a randomized, controlled trial, comparing treatment with an active control condition.

Hypothesis Primary hypothesis Patients with health anxiety treated with iACT will at 6-month follow-up report a significant reduction in illness worry compared to the action control condition iFORUM.

Secondary hypotheses

Patients with health anxiety treated with iACT compared to the active control condition iFORUM will at 6-month follow-up report:

1. a reduction in physical symptoms and symptoms of anxiety and depression
2. increased health-related quality of life
3. more expedient illness perceptions and increased acceptance of symptoms

   Mediation analyses
4. changes in illness perception and acceptance mediate the effect of iACT

ELIGIBILITY:
Inclusion Criteria:

1. Severe health anxiety > 6 months
2. Whiteley-7 score (scale 0-100 score points) corresponding to 21,4 or more.
3. Age above 18 years old
4. In case of a comorbid functional or other psychiatric disorder health anxiety must be the dominant problem
5. Patients who speak, read and write Danish
6. Access to a computer and internet access
7. Residence in Denmark

Exclusion criteria:

1. Acute suicidal risk
2. Abuse of narcotics or alcohol and (non-prescribed) medicine
3. Lifetime-diagnosis of psychoses, bipolar affective disorder or depression with psychotic symptoms (ICD-10: F20-29, F30-31, F32.3, F33.3)
4. Pregnancy
5. Unstable psychopharmacological treatment within last 2 months
6. Former treatment at the Research Clinic for Functional Disorders and Psychosomatics
7. Not providing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Whiteley-7 index | At baseline (i.e. at self-referral), before randomisation (i.e. after clinical assessment and up to 6 weeks after baseline) and 1, 2, 3 and 9 months after randomisation
  Health anxiety symptoms

SECONDARY OUTCOMES:
Demographic questions measured with questions from the Danish study for Functional Disorders (DanFund) | At baseline (i.e. at self-referral)
Diagnosed somatic illnesses measured with questions from the Danish study for Functional Disorders (DanFund) | At baseline (i.e. at self-referral)
Quality of life measured with the World Health Organisation Well-being Index-Five (WHO-5) | At baseline (i.e. at self-referral), before randomisation (i.e. after clinical assessment and up to 6 weeks after baseline) and 1, 2, 3 and 9 months after randomisation
Quality of life measured with the visual analogue scale (VAS question) from Youth profile, National Institute of Public Health | At baseline (i.e. at self-referral), before randomisation (i.e. after clinical assessment and up to 6 weeks after baseline) and 1, 2, 3 and 9 months after randomisation
Stress measured with questions from the survey Youth stress, Danish Health Authority | At baseline (i.e. at self-referral), before randomisation (i.e. after clinical assessment and up to 6 weeks after baseline) and 1, 2, 3 and 9 months after randomisation
Health anxiety symptoms measured with the Short Health Anxiety Inventory (SHAI) | At baseline (i.e. at self-referral), and 3 and 9 months after randomisation
Anxiety, depression, obsessive-compulsive and physical symptoms measured with subscales from the Symptom Checklist (SCL-92) | At baseline (i.e. at self-referral), and 3 and 9 months after randomisation
Somatisation measured with the Bodily Distress Syndrome Checklist (BDS Checklist) | At baseline (i.e. at self-referral)
General health status and functioning measured with the Short Form 12 Health Survey (SF-12) | At baseline (i.e. at self-referral), before randomisation (i.e. after clinical assessment and up to 6 weeks after baseline), 3 and 9 months after randomisation

OTHER OUTCOMES:
Psychological flexibility measured with the Acceptance and Action Questionnaire-II (AAQ-II) | At baseline (i.e. at self-referral), and 1, 2, 3 and 9 months after randomisation
Non-reactivity measured with a subscale of the Five Facet Mindfulness Questionnaire (FFMQ) | At baseline (i.e. at self-referral), and 1, 2, 3 and 9 months after randomisation
Illness perception measured with the Brief Illness Perception Questionnaire (B-IPQ) | At baseline (i.e. at self-referral), and 1, 2, 3 and 9 months after randomisation
Personality traits measured with the short version of the Big Five Inventory (BFI-10) | Before randomisation (i.e. after clinical assessment and up to 6 weeks after baseline)
Working alliance measured with the Working Alliance Inventory, Patient version (WAI-pt) | 2 weeks into treatment, and 3 months after randomisation
Treatment credibility and expectancy measured with the credibility/ expectancy questionnaire | Before randomisation (i.e. after clinical assessment and up to 6 weeks after baseline)
Childhood history questionnaire | Before randomisation (i.e. after clinical assessment and up to 6 weeks after baseline)
Traumatic events in childhood measured with the Childhood traumatic event scale | Before randomisation (i.e. after clinical assessment and up to 6 weeks after baseline)
Attachment style measured with the questionnaire: Experiences in close relationships - relationship structures (ECR-RS) | Before randomisation (i.e. after clinical assessment and up to 6 weeks after baseline)
Treatment evaluation of negative effects measured with the Inventory for the assessment of negative effects of psychotherapy (INEP) | 9 months after randomisation
Attitudes toward seeking professional help | At baseline (i.e. at self-referral) and at 3 months after randomisation
Self-reported health care use, work performance and work absence measured with Trimbos/ institute of Health Policy and Management (iMTA) questionnaire for Costs associated with Psychiatric Illness (TiC-P) | At baseline (i.e. at self-referral) and at 9 months after randomisation
Health care expenditures extracted from Danish national registers, and degree of illness related absence from work extracted from the Danish Register of Sickness absence compensation benefits and Social transfer payments database (DREAM). | At baseline (i.e. at self-referral) and at 9 months after randomisation
Health literacy measured with the Health Literacy Questionnaire (HLQ) | At baseline (i.e. at self-referral)
Values measured with the Sources of Meaning and Meaning in life questionnaire (SoMe-26) | At baseline (i.e. at self-referral), and 1, 2, 3 and 9 months after randomisation
Negative events and effects of psychological treatment | At 3 months after randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Lisbeth Frostholm, PhD, Principal Investigator — Aarhus University Hospital; Charlotte U Rask, PhD, Principal Investigator — Aarhus University Hospital

REFERENCES:
- [Derived] Risor BW, Frydendal DH, Villemoes MK, Nielsen CP, Rask CU, Frostholm L. Cost Effectiveness of Internet-Delivered Acceptance and Commitment Therapy for Patients with Severe Health Anxiety: A Randomised Controlled Trial. Pharmacoecon Open. 2022 Mar;6(2):179-192. doi: 10.1007/s41669-021-00319-x. Epub 2022 Jan 8. PMID 34997899
- [Derived] Hoffmann D, Rask CU, Hedman-Lagerlof E, Jensen JS, Frostholm L. Efficacy of internet-delivered acceptance and commitment therapy for severe health anxiety: results from a randomized, controlled trial. Psychol Med. 2021 Nov;51(15):2685-2695. doi: 10.1017/S0033291720001312. Epub 2020 May 14. PMID 32404226
- [Derived] Hoffmann D, Rask CU, Hedman-Lagerlof E, Eilenberg T, Frostholm L. Accuracy of self-referral in health anxiety: comparison of patients self-referring to internet-delivered treatment versus patients clinician-referred to face-to-face treatment. BJPsych Open. 2019 Sep 9;5(5):e80. doi: 10.1192/bjo.2019.54. PMID 31496462
- See also: Homepage for the Research Clinic for Functional Disorders, Aarhus University Hospital — http://www.functionaldisorders.dk